CLINICAL TRIAL: NCT00123994
Title: Tai Chi or Hydrotherapy for People With Osteoarthritis of the Hip(s) or Knee(s)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St George Hospital, Australia (Other)
Collaborators: Australian Government Department of Health and Ageing (Other Government); St George Division of General Practice, NSW, Australia. (Unknown); The University of New South Wales (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAMCIG56; RFP 95/0203
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2005-11-03 (Estimated); Status verified 2005-07

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: TaiChi; Hydrotherapy; Exercise; Joint pain; Disability
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Motor Activity; Arthralgia

INTERVENTIONS:
Behavioral: Tai Chi classes
Behavioral: Hydrotherapy classes

SUMMARY:
The aim of this study is to determine, in the framework of a randomized controlled clinical trial, whether Tai Chi can affect measurable improvements in self-reported outcomes such as pain, physical function and psychological well-being in people with osteoarthritis (OA) mainly affecting the hips or knees. The effectiveness of Tai Chi will be compared with both a non-intervention control group as well as with a formal exercise program, hydrotherapy. Hydrotherapy has long been considered an effective intervention for people with chronic OA although scientific evidence is weak at present. The main study hypotheses are that Tai Chi or hydrotherapy can significantly decrease pain and physical limitations; improve health-related quality of life; and promote psychological well being in patients with OA of the hip(s) or knee(s); and that Tai Chi and hydrotherapy are of equal efficacy.

DETAILED DESCRIPTION:
A single blinded randomized controlled clinical trial with 3 allocation groups:

* Tai Chi: maximum 15 people per group, twice weekly, 12 weeks.
* Hydrotherapy: maximum 15 people per group, twice weekly, 12 weeks.
* Control: 12 weeks waiting time prior to allocation to active intervention.

A specially designed Tai Chi program (Tai Chi for Arthritis, Paul Lam) will be provided in a community setting by trained instructors. Hydrotherapy sessions will be held at the St. George Hospital under supervision of registered physiotherapists with rheumatology and hydrotherapy experience.

Outcomes will be measured twice: 12 and 24 weeks after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the hip(s) or knee(s) according to American College of Rheumatology (ACR) clinical and radiographic (hip) criteria.

Exclusion Criteria:

* Currently participating in recreational physical activity more than twice a week.
* Unable to walk indoors for more than 10 minutes without a walking aid.
* Unable to exercise at a moderate level due to major co-morbidity.
* Incontinent, afraid of water or uncontrolled epilepsy.
* Low back pain referring to limbs.
* Joint replacement surgery in past year.
* Arthroscopic surgery or intra-articular injections in knee or hip in past 3 months.

Ages: 59 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-02; Study Completion 2005-10

PRIMARY OUTCOMES:
Self-reported pain and function (WOMAC)

SECONDARY OUTCOMES:
General health status (SF-36)
Psychological well being (DASS)
Patient global assessment (100mm visual analogue scale [VAS])
Physical performance: 50 feet walk time, stair time

CONTACTS AND LOCATIONS:
Overall Officials: Marlene H Fransen, PhD MPH, Principal Investigator — The George Institute, University of Sydney; John Edmonds, MB, BS, Study Chair — St George Hospital, University of NSW
Locations (1):
- St George Hospital, Kogarah, New South Wales, Australia

REFERENCES:
- [Derived] Fransen M, Nairn L, Winstanley J, Lam P, Edmonds J. Physical activity for osteoarthritis management: a randomized controlled clinical trial evaluating hydrotherapy or Tai Chi classes. Arthritis Rheum. 2007 Apr 15;57(3):407-14. doi: 10.1002/art.22621. PMID 17443749